CLINICAL TRIAL: NCT00012350
Title: Phase II Evaluation of FTI (R115777) (NSC 702818) in Treatment of Advanced Multiple Myeloma
Brief Title: Phase II Evaluation of FTase Inhibitor (FTI)in Treatment of Advanced Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-12516; NIH-2030 (Other: NIH); NCT00021203 (obsolete NCT alias)
Record Dates: First submitted 2001-03-03; First posted 2004-05-20 (Estimated); Last update posted 2012-10-23 (Estimated); Status verified 2012-10

CONDITIONS: Multiple Myeloma
Keywords: refractory multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; plasma cell neoplasm
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — tipifarnib; 2-(2-oxo-2-((3,7,11-trimethyl-2,6,10-dodecatrienyl)oxy)aminoethyl)phosphonic acid, (2,2-dimethyl-1-oxopropoxy)methyl ester sodium

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oral FTI (R115777) Treatment (Experimental): Patients will be administered oral FTI (R115777) at a dose of 300-mg by mouth (PO) twice a day (BID). Drug will be taken without regard to meals.
  The study regimen will consist of 3 weeks of treatment followed by one week off for a total cycle duration of 4 weeks.
  Interventions: Drug: FTI

INTERVENTIONS:
Drug: FTI
  Other Names: R115777; NSC702818; FTase Inhibitor; Tipifarnib; Zarnestra; farnesyl transferase inhibitor

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of R115777 in treating patients who have relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the rate of objective response and disease stabilization in patients with relapsed or refractory multiple myeloma treated with R115777. II. Determine whether the degree of inhibition of FTase activity and farnesylation of lamin-B, H-, K-, and N-RAS in peripheral blood mononuclear cells and tumor tissue correlates with tumor response in patients treated with this regimen. III. Determine whether the presence of activating RAS mutations in myeloma cells predicts treatment response in patients treated with this regimen. IV. Correlate R115777 plasma levels and RAS mutation status with tumor response in patients treated with this regimen.

OUTLINE: Patients receive oral R115777 twice daily on days 1-21. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity. Patients are followed for at least 30 days.

PROJECTED ACCRUAL: Approximately 12-42 patients will be accrued for this study within 25 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of relapsed or refractory multiple myeloma confirmed by the presence of the following: Bone marrow plasmacytosis with at least 10 percent plasma cells Sheets of plasma cells OR Biopsy-proven plasmacytoma Documentation of at least one of the following criteria: Serum myeloma (M)-protein component at least 1.0 g/dL by serum protein electrophoresis Urine M-protein excretion more than 200 mg/24 hours by urine protein electrophoresis Stage IIA or IIIA disease Measurable disease The following are not considered measurable disease: Lytic bone lesions Anemia Bone marrow plasmacytosis Beta-2 microglobulin in serum Previously treated with conventional chemotherapy Progressing or relapsing disease at time of study

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Eastern Cooperative Oncology Group (ECOG) 0-3 Life expectancy: More than 8 weeks Hematopoietic: Absolute neutrophil count at least 1,000/mm^3 Hepatic: aspartate aminotransferase (AST) or alanine transaminase (ALT) no greater than 2 times upper limit of normal (ULN) Bilirubin no greater than 2 mg/dL Renal: Creatinine no greater than 1.5 times ULN Calcium no greater than 12 mg/dL Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception Capable of swallowing intact study medication tablets No concurrent serious infection No grade 3 or greater peripheral neuropathy No life-threatening illness unrelated to tumor No other active or invasive cancer within the past 3 years except nonmelanoma skin cancer

PRIOR CONCURRENT THERAPY: Biologic therapy: Prior thalidomide allowed At least 14 days since prior immunologic agents No concurrent immunologic agents Chemotherapy: See Disease Characteristics At least 3 weeks since prior cytotoxic chemotherapy No other concurrent cytotoxic therapy Endocrine therapy: At least 14 days since prior high-dose corticosteroids No concurrent hormonal therapy No concurrent corticosteroids Radiotherapy: At least 3 weeks since prior radiotherapy and recovered No concurrent radiotherapy Surgery: Not specified Other: No other concurrent cancer therapy Concurrent pamidronate or other bisphosphonates allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2001-01; Primary Completion 2003-09 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | 26 months
  The primary end point of the study is to determine the rate of objective response and disease stabilization. Responses were to be defined according to modified Southwest Oncology Group (SWOG) criteria. Disease progression was defined as a 25% increase in the serum M-component confirmed by a second measurement obtained within 1 to 4 weeks of the first measurement, or an increase in the 24-hour urine M-component by more than 50%, confirmed by a second measurement. Other criteria for disease progression included the need to administer radiotherapy, new lytic bone lesions, enlargement of existing bone lesions, or new soft tissue plasmacytomas.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, M.D., Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States